CLINICAL TRIAL: NCT05791903
Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory on The Comfort, Satisfaction and Sleep Quality of Intensive Care Patients
Brief Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory on of Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ebubekir Kaplan, PhD student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ebkrkpln
Record Dates: First submitted 2023-03-07; First posted 2023-03-30 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Critical Care; Patient Satisfaction
Keywords: comfort; satisfaction; quality of sleep
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Experimental, randomised controlled, single-blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: randomized
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the application process, individuals in the experimental group will receive care based on Kolcaba's comfort theory and comfort behaviour checklist during their stay in the ICU.
  Interventions: Other: Nursing Care Based on Kolcaba's Comfort Theory
- Control Group (No Intervention): In this study, the control group will receive standard care.

INTERVENTIONS:
Other: Nursing Care Based on Kolcaba's Comfort Theory — Comfort-orientated care
  Arms: Experimental Group

SUMMARY:
Nurses aim to care for people who can no longer carry out their life activities and needs, and to ensure that they can continue to live their lives as well as possible. The aim is to improve the quality of life by making life more comfortable through care. Comfort in care means solving the patient's problems, being peaceful and content, and relieving pain/suffering. Kolcaba explained that comfort theory can be used as a guide to meet the comfort needs of individuals in the care process. The theory explains the concept of comfort as relaxation, refreshment and the ability to overcome problems (superiority). According to this theory, the nurse identifies the comfort needs of the patient and family and plans and implements interventions to meet these needs. There are no studies in the literature that have investigated the effect of nursing care based on Kolcaba's comfort theory on the comfort, satisfaction and sleep quality of ICU patients. The aim of this study is to determine the effect of nursing care based on Kolcaba's Comfort Theory on the comfort, satisfaction and sleep quality of ICU patients.

DETAILED DESCRIPTION:
The study is a randomised controlled experimental study to determine the effect of nursing care based on Kolcaba's comfort theory on comfort, care satisfaction and sleep quality of intensive care patients. Power analysis was used to determine the sample size of the study. As a result of the power analysis, it was determined that a total of 44 participants, 22 participants in each group, should be reached to achieve 80% power with an effect size of 0.87, a margin of error of 0.05% and a confidence interval of 0.95%. To increase the reliability of the study, a total of 80 participants, 40 in the intervention group and 40 in the control group, should be included in the study, taking into account data loss. In this study, the control group will receive standard care and the intervention group will receive care based on Kolcaba's comfort theory. Data will be collected using the General Comfort Scale, the Newcastle Satisfaction Scale, the Richard Campbell Sleep Scale and the Comfort Behaviours Checklist.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* 18 years of age or older,
* Being open to communication,
* Clear state of consciousness
* Staying in the intensive care unit for at least 24 hours

Exclusion Criteria:

* The patient is taking sedative medication
* Being diagnosed with a sleep disorder,
* The use of sleeping pills,
* Loss of hearing and/or vision
* Use of a hearing aid
* Dependence on mechanical ventilator
* illiteracy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
General Comfort Scale | 24 hours later
  The scale, which was developed by Katharine Kolcaba in 1992 in order to determine the comfort needs of individuals, to evaluate the nursing initiatives that can provide comfort and the increase in comfort, was adapted to Turkish society by Kuğuoğlu and Karabacak in 2004.The scale, which is a four-point Likert-type scale with 48 items, was created by guiding the taxonomic structure consisting of the theoretical components of comfort, including 3 levels and 4 dimensions. Level; While the dimension is evaluated as relief (16 items), relief (17 items) and overcoming the problems (15 items); It is evaluated in three parts: physical (12 items), psychospritual (13 items) and socio-cultural (10 items). Negative expressions in the scale are calculated by reverse coding during the evaluation phase. While the lowest total score that can be obtained from the scale is 48, the highest total score is 192.
Comfort Behaviors Checklist | 24 hours later
  The Comfort Behaviour Checklist was developed by Katharina Kolcaba in 1989. The checklist is completed by the observer when it is not possible for the person to complete the questionnaire. The Comfort Behaviour Checklist consists of 30 behavioural indicators. In addition to these, Kolcaba suggests that if the checklist is the only tool used to measure comfort, the individual should give a numerical score for pain and comfort so that comfort can be objectively assessed.
Richard-Campbell Sleep Scale | 24 hours later
  The scale was developed by Richards et al. (1987) to assess sleep quality in intensive care units (Richards, 1987; Richards et al., 2000). The RQAS includes six items (depth of sleep, time to fall asleep, frequency of awakening, duration of wakefulness, quality of sleep and ambient noise level). The scale score is evaluated with the sum of the first five items. A score of 25 and below indicates very poor sleep, while a minimum score of 76 and above indicates very good sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin ÖZAKGÜL, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Van yüzüncü yıl university, Van, Turkey (Türkiye)